CLINICAL TRIAL: NCT03956888
Title: The Effects of N-Acetylcysteine on Oxidative Stress Markers in Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: The Anti-oxidant Effects of N-Acetylcysteine in Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Siriraj Hospital (Other)
Responsible Party: Principal Investigator, Kittipong Maneechotesuwan, Professor, Siriraj Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: TH_IIS_NAC_2018
Record Dates: First submitted 2018-06-07; First posted 2019-05-21 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Acetylcysteine

STUDY DESIGN:
Intervention Model Description: Pre-post study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- N-acetylcysteine treatment (Experimental): All COPD patients will be treated with N-acetylcysteine at the dose of 1200 mg per day (600 mg three times a day) for 4 weeks in addition to their current COPD medications without other mucolytic agents
  Interventions: Drug: N-acetylcysteine

INTERVENTIONS:
Drug: N-acetylcysteine — All COPD patients will be treated with N-acetylcysteine at the dose of 1200 mg per day (600 mg three times a day) for 4 weeks in addition to their current COPD medications without other mucolytic agents

SUMMARY:
Chronic obstructive pulmonary disease (COPD) is a condition defined as a disease state characterized by airflow limitation that is not fully reversible. The airflow limitation is usually progressive and is associated with an abnormal inflammatory response of lungs to noxious particles or gases, primarily caused by cigarette smoking. The accelerated decline in lung function is closely associated with an increased number of neutrophils in the sputum and hence with higher level of airway inflammation. It becomes clear that the inflammatory process potentiates as COPD progresses and exerts damage which is irreversible. Oxidative stress is inextricably linked to the inflammatory response.

There is increasing evidence that an oxidant/antioxidant imbalance, in favor of oxidants, occurs in COPD.

NAC has been reported to reduce the viscosity of sputum in both cystic fibrosis and COPD, facilitating the removal of pulmonary secretions. Moreover, by maintaining the airway clearance, it prevents bacterial stimulation of mucin production and hence mucus hypersecretion.

The superiority of NAC over the other mucolytics may be in its anti-inflammatory and antioxidant properties and its mucolytic actions.

The aim of this study is to evaluate the effects of treatment with NAC long on oxidative stress marker change and also explore the effect of NAC to airway inflammatory, lung function test and CAT scores. Selected oxidative stress marker was defined as 8 - isoprostane, protein carbonyl, DNA damage.

ELIGIBILITY:
Inclusion Criteria:

* Eligible stable COPD patients who are currently treated with only short-acting bronchodilator (salbutamol or fenoterol/ipratropium bromide) or long-acting bronchodilator (LABA or LAMA) or inhaled corticosteroids/LABA
* Pre-bronchodilator FEV1 ≥ 80% and < 80% predicted
* Current or ex-smokers (≥ 10 pack year)

Exclusion Criteria:

* Concomitant with active and old pulmonary TB, lung cancer, bronchiectasis, lung fibrosis, destroyed lung and other malignancies
* Recent acute coronary syndrome (within 12 weeks)
* Cerebrovascular disease without neurological recovery
* Cognitive impairment
* Recent acute exacerbation of COPD (within 4 weeks)
* Recent respiratory viral infection (within 4 weeks)
* Could not provide adequate sputum specimens
* Develop worsening of COPD symptoms during sputum induction
* Could not provide informed consent

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
Level of 8 - isoprostane, MDA and DNA damage in sputum | 4 weeks
  To measure the different level of 8 - isoprostane, MDA and DNA damage in sputum before and after treated with NAC long in patients in this study, Reduce from first measurement.
  The level of 8 - isoprostane, MDA and DNA damage are reported according to ELISA based on the manufacturer's instructions.

SECONDARY OUTCOMES:
Percentage of Neutrophil in sputum | 4 weeks
  To measure the number of Neutrophil in sputum before and after treated with NAC long in patients in this study, Reduce from first measurement.
  Total cell counts are recorded with on a hemocytometer, using Kimura staining. Cell viability is determined by Trypan blue exclusion before cytospins were undertaken. The slides are stained with May-Grunwald-Giemsa stain and differential cell counts were made by a blinded observer. Four hundred inflammatory cells are counted on two slides for each sample in a blinded manner. Differential cell counts are expressed as the percentages of total Neutrophil will be reported.
  Samples with cell viability of greater than 70% and less than 30% squamous cell contamination are considered adequate for analysis.
FVC | 4 weeks
  To measure the FVC with Spirometry before and after treated with NAC long in patients in this study, improve from first measurement in FVC will be reported.
FEV1 | 4 weeks
  To measure the FEV1 with Spirometry before and after treated with NAC long in patients in this study, improve from first measurement in FEV1 will be reported.
FEV1/FVC | 4 weeks
  To measure the FEV1/FVC with Spirometry before and after treated with NAC long in patients in this study, improve from first measurement in FEV1/FVC will be reported.
COPD Assessment Test (CAT TM) | 4 weeks
  To measure the COPD Assessment Test (CATTM) before and after treated with NAC long in patients in this study.
  CATTM is Patient-completed questionnaire assessing globally the impact of COPD (cough, sputum, dyspnea, chest tightness) on health status of COPD patient.
  The minimum score is Zero (0) and the maximum score is Forty (40). Please see the correlation of score and impact level as in below table.
  CAT score
  Impact level
  >30 = Very high
  >20 = High
  10-20 = Medium
  <10 = Low
  5 = -
  In each question, there are score from 0 to five, the higher values represent the worse current situation. Score from each question will be summed then interpret based on CATTM Healthcare Professional User Guide ,Reduce test score from first measurement will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Kittipong Maneechotesuwan, MD., PhD., Principal Investigator — Siriraj Hospital
Locations (1):
- Faculty of Medicine, Siriraj Hospital, Mahidol University, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Undecided